CLINICAL TRIAL: NCT03157934
Title: Schlaganfallkonsortium Rhein-Neckar (Stroke Consortium Rhine-Neckar)
Acronym: FAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Dietmar Hopp Stiftung (Other)
Responsible Party: Principal Investigator, Prof. Dr. Wolfgang Wick, Chairman of the Neurologic Clinic, University Hospital Heidelberg
Other Study IDs: FAST
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Stroke; Vascular Diseases; Cardiovascular Diseases
Keywords: stroke network; acute stroke care; emergency medical services; integrated care
MeSH Terms: conditions — Ischemic Stroke; Vascular Diseases; Cardiovascular Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary CSC (Comprehensive Stroke center) admission: Patients with primary admission to endovascular-ready hospital (comprehensive stroke center)
  Interventions: Other: not applicable (observational study)
- Primary non-CSC (non-Comprehensive Stroke Center) SU (Stroke Unit) admission: Patients with primary admission to non-endovascular-ready hospital with (regional/local) stroke unit
  Interventions: Other: not applicable (observational study)
- Non-acute stroke hospital admission: Patients with primary admission to non-acute stroke-ready hospital
  Interventions: Other: not applicable (observational study)

INTERVENTIONS:
Other: not applicable (observational study) — Observational study without study related intervention

SUMMARY:
FAST is an investigator-initiated multicenter study embedded in a German multistate acute stroke network. The main objectives of the FAST study are to improve outcomes and quality of care for stroke patients, to quantify the number of patients in need of thrombectomy within an integrated stroke network, to study the best way of delivering and performing thrombectomy and to investigate the best model of pre-hospital selection and referral for stroke patients.

DETAILED DESCRIPTION:
Since 2015, mechanical thrombectomy in patients with large vessel occlusion has become an evidence based highly efficient treatment. In contrast to thrombolysis, thrombectomy can only be delivered by qualified interventionalists at comprehensive stroke centers. Thus, the implementation of thrombectomy into clinical practice remains a challenge. The investigators aim to establish a population based approach within a patient registry in a federal state overarching regional stroke network covering over 4 million inhabitants and integrating approximately 30 hospitals with different levels of expertise. The registry will include data from all acute ischemic stroke patients - approx. 12.000 patients p.a - within the network. The investigators plan to establish a central multi-interface platform integrating clinical data from the prehospital, intrahospital and rehabilitation phase including mandatory quality assurance, neurological and neuroradiological treatment and outcome data. The registry will allow addressing important questions, such as how many patients are candidates for thrombectomy, how many resources are needed to meet that demand and how treatment procedures and times can be improved. The overarching aim is to deliver high quality stroke care to every patient in the region.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients with ischemic stroke who are admitted to one of the hospitals of the Stroke Consortium Rhein-Neckar (FAST)
* informed consent

Exclusion Criteria:

* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute stroke patients admitted to one of the hospitals of the Stroke Consortium Rhein-Neckar (FAST)
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 3 months after intervention
  Functional outcome according to the modified Rankin Scale (mRS)

SECONDARY OUTCOMES:
Number of patients receiving acute recanalisation therapies of all referrals | 24 h after stroke onset
  Number of patients receiving thrombolysis and/or thrombectomy of all patients included in to the Network via the database.
Referral rates | Stroke onset to discharge from acute hospital; through study completion, an average of 2 years
  Referral rates by stroke service level (i.e. type of treatment center)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wick, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Heidelberg University Hospital, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Subject to approval by ethics committee

REFERENCES:
- See also: FAST on ResearchGate — https://www.researchgate.net/project/FAST-STROKE-CONSORTIUM-RHINE-NECKAR
- See also: FAST on Twitter — https://twitter.com/FAST_Heidelberg
- See also: FAST Website with download Resources — http://www.fast-schlaganfall.de